CLINICAL TRIAL: NCT03643003
Title: Music Therapy for Persons With Dementia: A Randomized Clinical Crossover Trial
Brief Title: Music Therapy for Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201709731
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Quality of Life; Social Interaction; Emotions; Mood; Feelings; Alzheimer Disease; Dementia
Keywords: music; music therapy
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Participants will engage in a music therapy condition of interest, and a non-music, verbal discussion comparison condition. The order is randomly assigned and counterbalanced across nursing homes, and all participants complete both conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): "Music therapy" consists of live singing of participant-preferred music, with guitar accompaniment, by a board-certified music therapist (i.e., MT-BC), following a protocol regarding how to manipulate the music in real time per participant responses. Order is randomly assigned, and all participants engage in both study arms.
  Interventions: Behavioral: Music therapy; Behavioral: Non-Music Verbal Interaction (Placebo)
- Non-Music Verbal Interaction (Placebo Comparator): "Non-music verbal interaction" consists of conversation of participants' interests, without music, by a board-certified music therapist, following a protocol regarding how to respond verbally in real time per participant responses. Order is randomly assigned, and all participants engage in both study arms.
  Interventions: Behavioral: Music therapy; Behavioral: Non-Music Verbal Interaction (Placebo)

INTERVENTIONS:
Behavioral: Music therapy — "Music therapy" consists of live singing of participant-preferred music, with guitar accompaniment, by a board-certified music therapist (i.e., MT-BC), following a protocol regarding how to manipulate the music in real time per participant responses. Dosage: participants engage in a small-group (3-6 participants) session at their nursing home, 3 times per week, across 2 consecutive weeks. Each session lasts 25 minutes and occurs in the afternoon.
Behavioral: Non-Music Verbal Interaction (Placebo) — "Non-music verbal interaction" consists of conversation of participants' interests, without music, by a board-certified music therapist, following a protocol regarding how to respond verbally in real time per participant responses. Dosage is the same as for music therapy: participants engage in a small-group (3-6 participants) session at their nursing home, 3 times per week, across 2 consecutive weeks. Each session lasts 25 minutes and occurs in the afternoon.

SUMMARY:
The purpose of this study is to examine the effectiveness of a specific, protocol-based group music therapy intervention, relative to a verbal discussion activity. The study will examine the impact of the specified music therapy intervention on: (1) affective outcomes, (2) social engagement behaviors, and (3) observed quality of life of persons with ADRD. This study will use a within-subjects randomized crossover design involving N=30 persons with ADRD from nursing homes to examine two levels of independent variable: singing-based music therapy and verbal discussion. Both conditions will be held in small groups of 3-6 participants. Nursing homes will be randomly assigned to an intervention sequence in a counterbalanced order (either music therapy first or verbal discussion first), and participants serve as their own controls. Each condition will occur three times per week for two consecutive weeks (6 sessions per treatment). Each session lasts for 25 minutes in the afternoon. A 2-week "wash-out" period (i.e., usual treatment) will occur between conditions. Participants will remain with their assigned small group for all study activities (i.e., music therapy, verbal discussion). Board-certified music therapists (i.e., MT-BC) will lead both conditions and will complete systematic training to ensure these conditions are implemented as intended, following a manualized protocol. An independent auditor will conduct random checks to ensure the music therapists are implementing the conditions as stipulated in the protocol. Data takers will complete systematic, manualized training to ensure reliable data collection.

DETAILED DESCRIPTION:
1. Following the consent process, the PI will collect demographics, music background, and preference information from participants' family and/or facility care staff. Where possible, the PI will ask participants directly about their music preferences.
2. The main study period will last 9 weeks and will consist of the following: (a) a "pre-study" week involving a practice session that includes aspects of both study conditions. All study personnel, and facility staff, will gain practice running through study procedures; (1) one week of usual treatment (UT) to collect baseline mood and quality of life data; (2-3) random assignment to two weeks of either music therapy or the verbal discussion; (4-5) a two-week washout period for collecting mood and quality of life data during return to UT; (6-7) crossover to the other condition; and (8) one final week return to UT with mood and quality of life data collection.
3. The PI will collect descriptive information during the pre-study week and first week of UT using the following measures (previously validated with this population):

   * Clinical Dementia Rating (CDR; Morris, 1993), consists of semi-structured interviews with the patient and an informant by a trained rater (in this case, the PI) regarding memory, orientation, judgment and problem solving, community affairs, hobbies, and personal care. Provides information depth. Scores range from 0 ("normal") to 3 (severe dementia).
   * Montreal Cognitive Assessment (MoCA; Nasreddine et al., 2005), a brief screening of cognitive function. Scores range from 0 (greatly impaired) to 30 (unimpaired). Provides a quick assessment of cognitive functioning.
   * Charlson Age-Comorbidity Index (CACI; Charlson et al., 1987), compares the severity of International Classification of Diseases diagnosis codes and provides a systematic way to quantify general health in clinical research, via chart review. Scores range from 0 (excellent health) to 37 (poor health).
   * Katz Index of Independence in Activities of Daily Living (Katz Index; Katz et al., 1970), a brief measure of basic daily functional activities. Scores range from 0 (total dependence) to 6 (independent).
4. Weekly measures (administered to facility care staff by data takers, or via REDCap, at the end of each of the 9 weeks of the study):

   * REDCap is a data management tool that provides a secure, reliable web-based interface for collecting, managing, and storing study information.
   * AD-RD Mood Scale: a proxy measure of mood (Tappen & Williams, 2008) that yields a positive mood total score with two subscores (spirited, contented) and a negative mood total score with three subscores (hostile, apathetic, sad).
   * QUALIDEM: a multidimensional proxy measure of quality of life that examines person-environment quality of life indicators that are specific to persons with ADRD (Ettema, 2007; Ettema at al., 2005).
5. Activity Involvement Checklist: A data taker will ask the activity directors at participating facilities to complete the Activity Checklist regarding the types of activities offered to participants in a typical week, and whether or not participants tend to join in these activities. Note that this tool will only be used once. The facility may also opt to complete this questionnaire electronically via REDCap.
6. Session measures, all administered by trained data takers during participation in either music therapy or verbal discussion:

   * Dementia Mood Picture Test (DMPT; Tappen & Barry, 1995), a 6-item self-report measure of participants' feelings using simple face drawings and verbal descriptors. Yields a single score that ranges from 0 (most negative mood) to 12 (most positive mood). Administered before and after each session.
   * Menorah Park Engagement Scale (MPES; Camp et al., 2015), an observational measure of social engagement and activity. Yields a profile of six engagement scores, averaged across 5-minute observation intervals. The MPES incorporate items from the Observed Emotion Rating Scale (OERS; Lawton et al., 1996; 1999), an observational measure of facial expressions that indicate basic emotions.
7. Session protocol (music therapy, verbal discussion): grounded in a conceptual framework based in extant literature regarding how the intervention is expected to influence affective, social, and quality of life outcomes. This framework consists of intervention strategies organized within 6 themes: cognition, attention, familiarity, audibility, structure, and autonomy. The music therapy condition consists of live singing with guitar accompaniment by a board-certified music therapist (i.e., MT-BC) using participant-preferred selections. The conceptual framework and accompanying strategies inform how the music is manipulated in real time by the music therapist to meet participants' momentary needs and demonstration of strengths. The verbal condition is designed as a non-music comparison using all of the same strategies and adaptations, but in a non-music context. It consists of live conversation led by an MT-BC using conversation starters centered around age-appropriate, familiar topics. For both condition, sessions will be centered around a main topic (Travel/Places, Nature/Hobbies, & Love/Friendship), each of which will be used in two consecutive sessions in the same order across all participants. Sessions will occur three times per week for two consecutive weeks (6 sessions per treatment). Each session lasts for 25 minutes in the afternoon.
8. "Pre-Study" Week: Practice session (one 30-minute session), the music therapist will practice aspects of both the music therapy protocol and the verbal discussion protocol. Data takers will practice all data collection procedures. Facility staff will gain practice transitioning participants to and from the sessions.
9. Week 1, UT (baseline; AD-RD Mood Scale, QUALIDEM).
10. Weeks 2-3, first randomly assigned condition - either music therapy first or verbal discussion first (DMPT pre/post session, MPES+OERS during session; AD-RD Mood Scale and QUALIDEM end-of-week)
11. Weeks 4-5, UT (washout/return to baseline; AD-RD Mood Scale, QUALIDEM).
12. Weeks 6-7, crossover to condition not yet received - either music therapy or verbal discussion (DMPT pre/post session, MPES+OERS during session; AD-RD Mood Scale and QUALIDEM end-of-week)
13. Week 8, UT (return to baseline; AD-RD Mood Scale, QUALIDEM).
14. Post-study: as a general measure of decline over the course of the study, the PI will re-administer the MoCA. To minimize burden on participants and nursing home staff, the PI will not re-administer any of the other pre-study assessments.

ELIGIBILITY:
Inclusion Criteria:

* Residents of nursing homes in Eastern Iowa
* Physician's diagnosis (e.g., primary care doctor, neurologist) of Alzheimer's disease (AD) or a related dementia (e.g., vascular)
* At least 65 years old
* English is first and primary language
* Have lived at facility for at least 3 months

Exclusion Criteria:

* Individuals who currently receive music therapy services from a board-certified music therapist
* Severe hearing loss that prohibits enjoyment of music
* Severe vision impairment that precludes seeing enlarged visual aids and font
* Those identified with "age-related cognitive decline" without a formal diagnosis of AD or a related dementia
* Individuals receiving hospice services or are bedridden
* Individuals with young onset AD
* Individuals with co-occurring Parkinson's disease, Huntington's disease, Down's syndrome, or severe mental illness (e.g., schizophrenia, bipolar disorder, major depressive or major anxiety disorder identified prior to dementia diagnosis)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Social Engagement Behavior Score | Week 8
  Refers to participants' involvement within the social environment, measured measured by trained data takers using the Menorah Park Engagement Scale (MPES; Camp et al., 2015). The MPES was designed for use with dementia patients. According to this scale, there are 5 categories of engagement: constructive, passive, other engagement, non-engagement, and disengagement. These categories are measured via behavioral observation in 5-minute observation intervals. Behaviors are rated: not at all (0), up to half of the observation interval (1 point), or more than half of the observation interval (2 points). The MPES incorporates the Observed Emotion Rating Scale, described in another section.
Emotion Behavior Score | Week 8
  Refers to participants' displayed facial expressions as an indicator of basic emotions, measured by trained data takers using the Observed Emotion Rating Scale (OERS; Lawton et al., 1996; 1999). The OERS was designed for use with dementia patients. Four of the 5 items on this scale will be used (pleasure, anger, anxiety/fear, depression/sadness; not interest) in 5-minute observation intervals during each session, in conjunction with the Menorah Park Engagement Scale (described in an earlier section).
Mood Behavior Score | Week 8
  Refers to behavioral indicators of emotion over a longer period of time (i.e., mood), measured using the AD-RD Mood Scale (Tappen & Williams, 2008; designed for use with dementia patients). This proxy measure will be completed weekly by facility care staff who have interacted frequently with participants over the past week. The scale yields a positive mood total score with two subscores (spirited, contented) and a negative mood total score with three subscores (hostile, apathetic, sad).
Self-Reported Feelings Score | Week 8
  Refers to momentary, self-reported feelings of participants before and after music therapy and verbal discussion sessions. Measured using the Dementia Mood Picture Test (DMPT; Tappen & Barry, 1995), which is a 6-item self-report measure that was designed to use with patients with more severe dementia. It uses simple face drawings and verbal descriptors to facilitate a response. Yields a single score that ranges from 0 (most negative mood) to 12 (most positive mood). Administered before and after each session.
Quality of Life Behavior Score | Week 8
  Refers to behavioral indicators of quality of life over a week, measured using the QUALIDEM (Ettema, 2007; Ettema at al., 2005; designed for use with dementia patients). This proxy measure will be completed weekly by facility care staff who have interacted frequently with participants over the past week. This measure considers multiple person-environment dimensions of how the individual with dementia interacts with his or her environment, and includes objective environmental and behavioral components, the patient's subjective experience, and how the person functions within the social environment.

CONTACTS AND LOCATIONS:
Overall Officials: Alaine Reschke-Hernandez, MA, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen-Mansfield J, Dakheel-Ali M, Marx MS. Engagement in persons with dementia: the concept and its measurement. Am J Geriatr Psychiatry. 2009 Apr;17(4):299-307. doi: 10.1097/JGP.0b013e31818f3a52. PMID 19307858
- [Background] Cohen-Mansfield J, Marx MS, Freedman LS, Murad H, Regier NG, Thein K, Dakheel-Ali M. The comprehensive process model of engagement. Am J Geriatr Psychiatry. 2011 Oct;19(10):859-70. doi: 10.1097/JGP.0b013e318202bf5b. PMID 21946802
- [Background] Feinstein JS, Duff MC, Tranel D. Sustained experience of emotion after loss of memory in patients with amnesia. Proc Natl Acad Sci U S A. 2010 Apr 27;107(17):7674-9. doi: 10.1073/pnas.0914054107. Epub 2010 Apr 12. PMID 20385824
- [Background] Ferguson SH, Quene H. Acoustic correlates of vowel intelligibility in clear and conversational speech for young normal-hearing and elderly hearing-impaired listeners. J Acoust Soc Am. 2014 Jun;135(6):3570-84. doi: 10.1121/1.4874596. PMID 24907820
- [Background] Hebert LE, Weuve J, Scherr PA, Evans DA. Alzheimer disease in the United States (2010-2050) estimated using the 2010 census. Neurology. 2013 May 7;80(19):1778-83. doi: 10.1212/WNL.0b013e31828726f5. Epub 2013 Feb 6. PMID 23390181
- [Background] Janata P. The neural architecture of music-evoked autobiographical memories. Cereb Cortex. 2009 Nov;19(11):2579-94. doi: 10.1093/cercor/bhp008. Epub 2009 Feb 24. PMID 19240137
- [Background] Keeler JR, Roth EA, Neuser BL, Spitsbergen JM, Waters DJ, Vianney JM. The neurochemistry and social flow of singing: bonding and oxytocin. Front Hum Neurosci. 2015 Sep 23;9:518. doi: 10.3389/fnhum.2015.00518. eCollection 2015. PMID 26441614
- [Background] Koelsch S. Toward a neural basis of music perception - a review and updated model. Front Psychol. 2011 Jun 9;2:110. doi: 10.3389/fpsyg.2011.00110. eCollection 2011. PMID 21713060
- [Background] Kolanowski A, Litaker M, Buettner L, Moeller J, Costa PT Jr. A randomized clinical trial of theory-based activities for the behavioral symptoms of dementia in nursing home residents. J Am Geriatr Soc. 2011 Jun;59(6):1032-41. doi: 10.1111/j.1532-5415.2011.03449.x. Epub 2011 Jun 7. PMID 21649633
- [Background] Kverno KS, Black BS, Nolan MT, Rabins PV. Research on treating neuropsychiatric symptoms of advanced dementia with non-pharmacological strategies, 1998-2008: a systematic literature review. Int Psychogeriatr. 2009 Oct;21(5):825-43. doi: 10.1017/S1041610209990196. Epub 2009 Jul 9. PMID 19586562
- [Background] Livingston G, Kelly L, Lewis-Holmes E, Baio G, Morris S, Patel N, Omar RZ, Katona C, Cooper C. A systematic review of the clinical effectiveness and cost-effectiveness of sensory, psychological and behavioural interventions for managing agitation in older adults with dementia. Health Technol Assess. 2014 Jun;18(39):1-226, v-vi. doi: 10.3310/hta18390. PMID 24947468
- [Background] McDermott O, Orrell M, Ridder HM. The importance of music for people with dementia: the perspectives of people with dementia, family carers, staff and music therapists. Aging Ment Health. 2014;18(6):706-16. doi: 10.1080/13607863.2013.875124. Epub 2014 Jan 13. PMID 24410398
- [Background] Millan-Calenti JC, Lorenzo-Lopez L, Alonso-Bua B, de Labra C, Gonzalez-Abraldes I, Maseda A. Optimal nonpharmacological management of agitation in Alzheimer's disease: challenges and solutions. Clin Interv Aging. 2016 Feb 22;11:175-84. doi: 10.2147/CIA.S69484. eCollection 2016. PMID 26955265
- [Background] Muller V, Lindenberger U. Cardiac and respiratory patterns synchronize between persons during choir singing. PLoS One. 2011;6(9):e24893. doi: 10.1371/journal.pone.0024893. Epub 2011 Sep 21. PMID 21957466
- [Background] Osman SE, Tischler V, Schneider J. 'Singing for the Brain': A qualitative study exploring the health and well-being benefits of singing for people with dementia and their carers. Dementia (London). 2016 Nov;15(6):1326-1339. doi: 10.1177/1471301214556291. Epub 2014 Nov 24. PMID 25425445
- [Background] Reschke-Hernandez AE, Okerstrom KL, Bowles Edwards A, Tranel D. Sex and stress: Men and women show different cortisol responses to psychological stress induced by the Trier social stress test and the Iowa singing social stress test. J Neurosci Res. 2017 Jan 2;95(1-2):106-114. doi: 10.1002/jnr.23851. PMID 27870432
- [Background] Sakamoto M, Ando H, Tsutou A. Comparing the effects of different individualized music interventions for elderly individuals with severe dementia. Int Psychogeriatr. 2013 May;25(5):775-84. doi: 10.1017/S1041610212002256. Epub 2013 Jan 8. PMID 23298693
- [Background] Schubert E. Emotion felt by the listener and expressed by the music: literature review and theoretical perspectives. Front Psychol. 2013 Dec 17;4:837. doi: 10.3389/fpsyg.2013.00837. PMID 24381565
- [Background] Tappen RM, Williams CL. Development and testing of the Alzheimer's Disease and Related Dementias Mood Scale. Nurs Res. 2008 Nov-Dec;57(6):426-35. doi: 10.1097/NNR.0b013e31818c3dcc. PMID 19018217
- [Background] Witek MA, Clarke EF, Wallentin M, Kringelbach ML, Vuust P. Syncopation, body-movement and pleasure in groove music. PLoS One. 2014 Apr 16;9(4):e94446. doi: 10.1371/journal.pone.0094446. eCollection 2014. PMID 24740381
- [Background] Beerens HC, Zwakhalen SM, Verbeek H, Ruwaard D, Hamers JP. Factors associated with quality of life of people with dementia in long-term care facilities: a systematic review. Int J Nurs Stud. 2013 Sep;50(9):1259-70. doi: 10.1016/j.ijnurstu.2013.02.005. Epub 2013 Mar 5. PMID 23465959
- [Background] Blackburn R, Bradshaw T. Music therapy for service users with dementia: a critical review of the literature. J Psychiatr Ment Health Nurs. 2014 Dec;21(10):879-88. doi: 10.1111/jpm.12165. Epub 2014 Oct 10. PMID 25303405
- [Background] Brasure M, Jutkowitz E, Fuchs E, Nelson VA, Kane RA, Shippee T, Fink HA, Sylvanus T, Ouellette J, Butler M, Kane RL. Nonpharmacologic Interventions for Agitation and Aggression in Dementia [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2016 Mar. Report No.: 16-EHC019-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK356163/ PMID 27099894
- [Background] Guzman-Velez E, Feinstein JS, Tranel D. Feelings without memory in Alzheimer disease. Cogn Behav Neurol. 2014 Sep;27(3):117-29. doi: 10.1097/WNN.0000000000000020. PMID 25237742
- [Background] Juslin PN. From everyday emotions to aesthetic emotions: towards a unified theory of musical emotions. Phys Life Rev. 2013 Sep;10(3):235-66. doi: 10.1016/j.plrev.2013.05.008. Epub 2013 May 29. PMID 23769678
- [Background] Robb SL, Burns DS, Carpenter JS. Reporting Guidelines for Music-based Interventions. Music Med. 2011 Oct;3(4):271-279. doi: 10.1177/1943862111420539. PMID 23646227
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Numminen A, Kurki M, Johnson JK, Rantanen P. Cognitive, emotional, and social benefits of regular musical activities in early dementia: randomized controlled study. Gerontologist. 2014 Aug;54(4):634-50. doi: 10.1093/geront/gnt100. Epub 2013 Sep 5. PMID 24009169
- [Background] Tappen RM, Barry C. Assessment of affect in advanced Alzheimer's disease: the Dementia Mood Picture Test. J Gerontol Nurs. 1995 Mar;21(3):44-6. doi: 10.3928/0098-9134-19950301-09. No abstract available. PMID 7706649
- [Background] van der Steen JT, van Soest-Poortvliet MC, van der Wouden JC, Bruinsma MS, Scholten RJ, Vink AC. Music-based therapeutic interventions for people with dementia. Cochrane Database Syst Rev. 2017 May 2;5(5):CD003477. doi: 10.1002/14651858.CD003477.pub3. PMID 28462986
- [Background] Ettema TP, Droes RM, de Lange J, Ooms ME, Mellenbergh GJ, Ribbe MW. The concept of quality of life in dementia in the different stages of the disease. Int Psychogeriatr. 2005 Sep;17(3):353-70. doi: 10.1017/s1041610205002073. PMID 16252370
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Background] Katz S, Downs TD, Cash HR, Grotz RC. Progress in development of the index of ADL. Gerontologist. 1970 Spring;10(1):20-30. doi: 10.1093/geront/10.1_part_1.20. No abstract available. PMID 5420677
- [Background] van der Ploeg ES, Eppingstall B, Camp CJ, Runci SJ, Taffe J, O'Connor DW. A randomized crossover trial to study the effect of personalized, one-to-one interaction using Montessori-based activities on agitation, affect, and engagement in nursing home residents with Dementia. Int Psychogeriatr. 2013 Apr;25(4):565-75. doi: 10.1017/S1041610212002128. Epub 2012 Dec 14. PMID 23237211
- See also: Alzheimer's Association — http://www.alz.org/facts/overview.asp
- See also: American Music Therapy Association — http://www.musictherapy.org